CLINICAL TRIAL: NCT01331928
Title: A Phase II Study of Sequential Capecitabine Plus Oxaliplatin (XELOX) Followed by Docetaxel Plus Capecitabine (TX) in Patients With Unresectable Gastric
Brief Title: Sequential Chemotherapy With Xelox Follows by TX to Treat Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Chao Yee, Taipei Veterans General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOH99-TD-C-111-007
Record Dates: First submitted 2011-02-15; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-01

CONDITIONS: Gastric Cancer
Keywords: Sequential chemotherapy, gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine, Oxaliplatin, Docetaxel , Gastric cancer (Experimental)
  Interventions: Drug: Capecitabine (Xeloda, Roche), Oxaliplatin (Sanofi-Aventis), Docetaxel (Sanofi-Aventis)

INTERVENTIONS:
Drug: Capecitabine (Xeloda, Roche), Oxaliplatin (Sanofi-Aventis), Docetaxel (Sanofi-Aventis) — capecitabine orally 1000 mg/m2 twice daily, day1 to day 10, every 2 weeks plus oxaliplatin 85mg/m2 (2hrs IV infusion)on day1, every 2 weeks for 6 cycles, then shift to docetaxel 30 mg/m2(over 30-minute intravenous infusion) on day 1 and day 8 plus oral capecitabine 825 mg/m2 twice daily on day 1 to 14, every 3 weeks for 4 cycles.

SUMMARY:
The purpose of this study is to determine whether sequential chemotherapy with capecitabine plus oxaliplatin (Xelox) followed by docetaxel plus capecitabine (TX)in unresectable gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is one of the most frequent cancer types in Taiwan. Advanced gastric cancer is incurable. Although chemotherapy can improve survival and maintain quality of life for patients with advanced gastric cancer, optimal chemotherapy for this disease has not been defined.

Cytotoxic agents commonly used in this disease include platinum compounds, fluoropyrimidines and taxanes. A phase III (V325) study showed that adding docetaxel to cisplatin and 5-FU (TCF) improved response rates, progression-free survival (PFS), and overall survival (OS). Although the TCF regimen improved clinical outcomes, it was associated with substantial toxicity particularly that related to myelosuppression, with a 29% incidence of febrile neutropenia or neutropenic infection1. Several modifications to the TCF regimen have been made to maintain efficacy and reduce toxicity.

Cunningham et al. evaluated the impact of substituting oxaliplatin for cisplatin and capecitabine for 5-FU in the epirubicin, cisplatin, and 5-FU (ECF) regimen. Oxaliplatin as compared with cisplatin demonstrated comparable efficacy, with a lower incidence of myelosuppression, thromboembolic complications, and nephrotoxicity. The combination of docetaxel and oxaliplatin has been evaluated in gastric cancer with moderate activities in four phase II trials.

A different way of including all active agents in the first line treatment of advanced gastric cancer is to use them sequentially. Sequential schedules may maximize the dose-intensity of each single agent and avoid the overlapping toxicity caused by the concomitant administration of active drugs. Two studies using sequential strategy to treat advanced gastric cancer were reported.7-8 One used docetaxel after PELF regimen, the other used cisplatin plus 5-Fluorouracil / leucovorin (5-FU/LV) followed by irinotecan plus 5-FU/LV, followed by docetaxel plus 5-FU/LV. Both studies shown that sequential approach produced a good treatment efficacy with manageable toxicities in the management of advanced gastric cancer.

In our hospital, we had completed two phase II studies in advanced gastric cancer, including XELOX (capecitabine plus oxaliplatin) and a modified TCF regimen (docetaxel plus cisplatin and oral tegafur/uracil plus leucovorin). After analyzing these results, the median time to response, time to progression and overall survival were around 3, 6, and 10 months, respectively. Overall response rate was around 50% for each.

Based on the above considerations and our previous experiences, we hence initiate this phase II study to evaluate the feasibility and the anti-tumor activity of a new strategy consists of two sequential regimens involving XELOX and TX in unresectable gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed gastric adenocarcinoma.
* At least one measurable lesion in a non-irradiated area.
* No prior exposure to systemic chemotherapy for advanced gastric cancer.
* For those have adjuvant chemotherapy after a curative gastrectomy, the last dosing of previous adjuvant chemotherapy should be at least 6 months before the start of this treatment.
* Aged > 20 years old.
* ECOG Performance Status <= 2.
* Life expectancy greater than 12 weeks.
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function

Exclusion Criteria:

* Patient who are receiving concurrent radiotherapy, chemotherapy or other experimental therapy. (Previous radiotherapy is allowable if the last dose was given more than 1 month before the protocol treatment).
* Major surgery within two weeks prior to entering the study.
* Patients with CNS metastasis, including clinical suspicion.
* Patients who are under active or uncontrolled infections.
* Patients who had cardiac arrhythmia or myocardial infarction history 6 months before entry.
* Patients with clinically detectable peripheral neuropathy > 2 on the CTC criteria
* Patients with concomitant illness that might be aggravated by chemotherapy.
* Patients who are pregnant or with breast feeding.
* Other concomitant or previously malignancy within 5 yrs except for in situ cervix cancer or squamous cell carcinoma of the skin treated by surgery only.
* Patients with hypersensitivity to any component of the chemotherapeutic regimen.
* mental status is not fit for clinical trial
* can not take study medication orally
* fertile men and women unless using a reliable and appropriate contraceptive method

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
objective tumor response rate | 2 year
  Analysis for the objective response rate will be conducted on both the intention-to-treat (ITT) and evaluable data sets. Response will be assessed by Response Evaluation Criteria in Solid Tumor (RECIST 1.1).The analysis will be in descriptive statistics, presented by point estimate and 95% confidence interval for the efficacy variable (Objective tumor response rate)

SECONDARY OUTCOMES:
the progression-free survival, overall survival, toxicity profiles | 2 year
  The progression-free survival is defined as the duration between the time from the date of randomization to the date of first observed progressive disease or death due to any cause. The overall survival is defined as the duration between the time from the date of randomization to the date of death due to any cause.
  Toxicity profiles: measure numbers of participants with adverse events. Treatment toxicity will be graded by NCI Common Toxicity Criteria Version 4.0 (CTC,v4.0) for safety evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Chao, MD,PHD, Principal Investigator — attending physician, cancer center, Taipei Veterans General Hospital
Locations (1):
- Taipei veterans general hospital, Taipei, Taiwan, Taiwan